CLINICAL TRIAL: NCT04119674
Title: Pilot Study of Anlotinib in Combination With STUPP Regimen for Treatment of Patients With Newly Diagnosed Glioblastoma
Brief Title: Pilot Study of Anlotinib With STUPP Regimen for Patients With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen yuanyuan, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBM-AS
Record Dates: First submitted 2019-10-06; First posted 2019-10-08 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm (Experimental): single-arm Drug: Anlotinib Drug: Temozolomide Radiotherapy:Radiotherapy was initiated 4 to 6 weeks postoperatively at a dose of 1.8-2.0 Grays (Gy) per fraction for 5 days per week for 6 weeks with a total dose of 54-60 Gy.
  Interventions: Drug: Drug is Anlotinib.; Drug: Drug is Temozolomide Capsule.; Radiation: Radiotherapy was initiated 4 to 6 weeks postoperatively.

INTERVENTIONS:
Drug: Drug is Anlotinib. — Anlotinib 8 mg/day (Chia-tai Tianqing Pharmaceutical Co., Ltd.) was given orally on days 1 to 14 per 3-week cycle for 2 cycles during concomitant therapy and maximally 8 cycles during adjuvant chemotherapy. One week after discontinuation of adjuvant chemotherapy, anlotinib 8 mg/day was given for maintenance .
Drug: Drug is Temozolomide Capsule. — Temozolomide 75 mg/m2/day was taken for maximally 49 days during concurrent chemoradiotherapy. Beginning 4 weeks after completion of concurrent chemoradiotherapy, patients received adjuvant temozolomide for 5 days every 28 days, first cycle 150 mg/m2/day and subsequent cycles 200 mg/m2/day for maximally 6 cycles .
Radiation: Radiotherapy was initiated 4 to 6 weeks postoperatively. — Radiotherapy was initiated 4 to 6 weeks postoperatively at a dose of 1.8-2.0 Grays (Gy) per fraction for 5 days per week for 6 weeks with a total dose of 54-60 Gy.

SUMMARY:
The purpose of this study is to test the the efficacy and safety of Anlotinib in combination with STUPP regimen for patients with newly diagnosed glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Primary, pathologically confirmed glioblastoma, and complete molecular biological marker tests (MGMT, 1p/19q, IDH, TERT, BRAF, p53, EGFR);
2. 2 ~ 6 weeks after operation; the surgical incision healed well;
3. Presence of lesions evaluable according to Rano criteria;
4. Aged 18-70 years;
5. Karnofsky performance status (KPS) ≥ 60;
6. The dose of corticosteroid therapy was stable or gradually reduced in the past 5 days;
7. No previous radiotherapy, chemotherapy, immunotherapy, or biologic therapy;
8. Serum hemoglobin ≥ 100 g/L, platelet count ≥ 80 × 109/L, neutrophil count ≥ 1.5 × 109/L;
9. Serum creatinine ≤ 1.25 × ULN or creatinine clearance ≥ 60 mL/min;
10. Serum bilirubin ≤ 1.5 × ULN, AST (SGOT) and ALT (SGPT) ≤ 2.5 × ULN, alkaline phosphatase ≤ 5 × ULN;
11. Normal coagulation function (PT prolongation does not exceed 3s, APTT prolongation does not exceed 10s);
12. Women of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days prior to enrollment and be willing to use an appropriate method of contraception during the trial and 8 days after administration of the trial drug. Males must agree to use an appropriate method of contraception or be surgically sterile during the trial and after 8 weeks of trial drug administration;
13. Patient is sufficiently compliant with study and follow-up procedures;
14. Patients signed a formal informed consent form to indicate that they understood that the study was in accordance with hospital policy and ethical requirements.

Exclusion Criteria:

1. Secondary glioblastoma;
2. Patients with any other malignant tumor before or now, except skin non-melanotic carcinoma or cervical carcinoma in situ;
3. Any other diseases or conditions are contraindications to chemoradiotherapy (such as active phase of infection, within 6 months after cerebral myocardial infarction, symptomatic heart disease including unstable angina pectoris, congestive heart failure or uncontrolled arrhythmia, immunosuppressive therapy);
4. Pregnant or lactating women;
5. Women and men who are likely to become pregnant but are unwilling to take appropriate contraceptive measures;
6. Evidence of hereditary bleeding constitution or coagulation disorders;
7. Patients requiring anticoagulant therapy due to other diseases;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
PFS | from enrollment to progression or death (for any reason),assessed up to 18months
  Progression-Free Survival

SECONDARY OUTCOMES:
OS | from enrollment to death (for any reason).assessed up to 24 months
  Overall Survival
adverse event | from enrollment to death (for any reason).assessed up to 24 months
  Adverse events are described in terms of CTC AE 5.0
Health-related quality of life | from enrollment to death (for any reason).assessed up to 24 months
  Health-related quality of life are measured by the EORTC-QL30/BN20.
Neurocognitive function | from enrollment to death (for any reason).assessed up to 24 months
  Neurocognitive function are measured by John-Hopkins adapted cognitive exam (ACE).

CONTACTS AND LOCATIONS:
Overall Officials: Chen Ming, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang cancer hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No